CLINICAL TRIAL: NCT03374020
Title: Retinal Imaging Using NOTAL-OCT
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: BNZ-0077-017
Record Dates: First submitted 2017-09-11; First posted 2017-12-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Age-Related Macular Degeneration; Diabetic Retinopathy
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intermediate AMD
  Interventions: Device: Notal OCT
- Advanced AMD
  Interventions: Device: Notal OCT
- DR without macular edema
  Interventions: Device: Notal OCT
- DR with macular edema
  Interventions: Device: Notal OCT

INTERVENTIONS:
Device: Notal OCT — Imaging using Notal OCT

SUMMARY:
Comparison between retinal measurements, done by the Notal-OCT imaging and a commercial OCT (Optical Coherence Tomography)

ELIGIBILITY:
Inclusion Criteria:

1. Ability and agreement to give informed consent (IC)
2. Diagnosis of AMD or DR in SE by OCT
3. Ability to undergo OCT scans
4. VA of 20/160 or better in SE

Exclusion Criteria:

1. AMD and DR in the same SE
2. Evidence of macular disease other than AMD or DME in SE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. AMD population - intermediate and advanced AMD (with active and non-active CNV)
  2. DR population. Patient with and without DME
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The level of agreement between NOTAL-OCT and commercial OCT in detecting fluid in the 10 central degrees of the macula. | 1 year
  OCT B-scans from both devices will be graded for fluid by an eye care professional and results per macula will be analyzed. A binary decision "there is fluid" or "there is no fluid" will be given to each macula (10 central degrees). Then agreement between decisions, commercial and Notal OCT, will be compared